CLINICAL TRIAL: NCT04017832
Title: China Multi-regional Clinical Trial: Efficacy and Safety of Oral Semaglutide Versus Sitagliptin in Subjects With Type 2 Diabetes Mellitus Treated With Metformin
Brief Title: A Research Study Comparing a New Medicine Oral Semaglutide to Sitagliptin in People With Type 2 Diabetes
Acronym: PIONEER 12
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9924-4309; U1111-1188-1256 (Other: World Health Organization (WHO)); 2018-002589-38 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2019-07-11; First posted 2019-07-12 (Actual); Results first posted 2023-09-29 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oral semaglutide 3 mg and placebo (sitagliptin) (Experimental): Oral semaglutide tablets 3 mg and sitagliptin placebo tablets for 26 weeks
  Interventions: Drug: Oral semaglutide; Drug: Placebo (sitagliptin)
- Oral semaglutide 7 mg and placebo (sitagliptin) (Experimental): Oral semaglutide tablets and sitagliptin placebo tablets. The dose of oral semaglutide will be escalated over 4 weeks, after which the target dose of 7 mg is taken for 22 weeks
  Interventions: Drug: Oral semaglutide; Drug: Placebo (sitagliptin)
- Oral semaglutide 14 mg and placebo (sitagliptin) (Experimental): Oral semaglutide tablets and sitagliptin placebo tablets. The dose of oral semaglutide will be escalated over 8 weeks, after which the target dose of 14 mg is taken for 18 weeks
  Interventions: Drug: Oral semaglutide; Drug: Placebo (sitagliptin)
- Sitagliptin 100 mg and placebo (oral semaglutide) (Experimental): Sitagliptin tablets and oral semaglutide placebo tablets for 26 weeks
  Interventions: Drug: Sitagliptin; Drug: Placebo (oral semaglutide)

INTERVENTIONS:
Drug: Oral semaglutide — Oral semaglutide to be taken every morning in a fasting state, to be followed by sitagliptin placebo after 30 minutes. Only then participants can have their first meal of the day and their pre-study metformin tablets
  Arms: Oral semaglutide 14 mg and placebo (sitagliptin); Oral semaglutide 3 mg and placebo (sitagliptin); Oral semaglutide 7 mg and placebo (sitagliptin)
Drug: Sitagliptin — Sitagliptin to be taken every morning, 30 minutes after taking the oral semaglutide placebo tablet. Then participants can have their first meal of the day and their pre-study metformin tablets
  Arms: Sitagliptin 100 mg and placebo (oral semaglutide)
Drug: Placebo (oral semaglutide) — Placebo tablet to be taken first thing in the morning
  Arms: Sitagliptin 100 mg and placebo (oral semaglutide)
Drug: Placebo (sitagliptin) — Placebo tablet to be taken 30 minutes after oral semaglutide
  Arms: Oral semaglutide 14 mg and placebo (sitagliptin); Oral semaglutide 3 mg and placebo (sitagliptin); Oral semaglutide 7 mg and placebo (sitagliptin)

SUMMARY:
This study compares 2 medicines for type 2 diabetes: oral semaglutide (a new medicine) and sitagliptin (a medicine doctors can already prescribe). Participants will either get oral semaglutide or sitagliptin - which treatment is decided by chance. Participants will get 2 tablets a day to take first thing in the morning on an empty stomach. Only 1 tablet has study medicine in it. The other tablet is a dummy medicine (placebo). After taking the semaglutide tablet, participants may not eat or drink anything for at least 30 minutes. After the 30 minutes, participants must take the sitagliptin tablet. Then participants can have their first meal of the day and take any other medicines they may need, including their metformin. The study will last for about 7 months (33 weeks). Participants will have 8 clinic visits and 1 phone call with the study doctor. At all 8 of the clinic visits, participants will have blood samples taken.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
* Male or female, age above or equal to 18 years at the time of signing informed consent.

For Algeria only: Male or female, age above or equal to 19 years at the time of signing informed consent.

For Taiwan only: Male or female, age above or equal to 20 years at the time of signing informed consent

* Diagnosed with type 2 diabetes mellitus 60 days or more prior to day of screening.
* HbA1c between 7.0-10.5% (53-91 mmol/mol) (both inclusive).
* Stable daily dose of metformin (equal to or above 1500 mg or maximum tolerated dose as documented in the subject medical record) 60 days or more prior to day of screening

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method (adequate contraceptive measure as required by local regulation or practice).
* Family or personal history of multiple endocrine neoplasia type 2 (MEN 2) or medullary thyroid carcinoma (MTC). Family is defined as a first degree relative.
* History or presence of pancreatitis (acute or chronic).
* History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery).
* Any of the following: myocardial infarction, stroke, hospitalization for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening and randomisation.
* Subjects presently classified as being in New York Heart Association (NYHA) Class IV.
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening.
* Renal impairment measured as estimated glomerular filtration rate (eGFR) below 60 mL/min/1.73 m^2 as per Chronic Kidney Disease Epidemiology Collaboration formula (CKD-EPI).
* Subjects with alanine aminotransferase (ALT) above 2.5 x upper limit of the normal (ULN).
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a pharmacologically pupil-dilated fundus examination performed by an ophthalmologist or another suitably qualified health care provider within the past 90 days prior to screening or in the period between screening and randomisation. Fundus examination without dilation is only allowed if the digital camera used for fundus photography has this feature.
* Presence or history of malignant neoplasms within the past 5 years prior to the day of screening. Basal and squamous cell skin cancer and any carcinoma in-situ is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1441 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (93):
- Algeria (2):
  - Maison des diabétiques El Harrach, Algiers
  - Department of internal medicine hospital (CHU) of BIRTRARIA, Algiers
- Brazil (3):
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul Ltda., Porto Alegre, Rio Grande do Sul
  - CPQuali Pesquisa Clínica Ltda, São Paulo, São Paulo
  - CPCLIN - Centro de Pesquisas Clínicas, São Paulo, São Paulo
- China (59):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Beijing Pinggu Hospital, Beijing, Beijing Municipality
  - Second Affliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - 900th Hospital of Joint Logistics Support Force, Fuzhou, Fujian
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - Shunde Hospital of Southern Medical University, Foshan, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen Universtiy, Guangzhou, Guangdong
  - Guangzhou Panyu Central Hospital, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - The 2nd Affiliated Hospital of Shantou Uni Medical College, Shantou, Guangdong
  - Cangzhou People's Hospital, Cangzhou, Hebei
  - Harrison International Peace Hospital, Hengshui, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - The First Affiliated Hospital of Henan university of Science, Luoyang, Henan
  - Zhengzhou First People's Hospital, Zhengzhou, Henan
  - Taihe Hospital, Shiyan, Hubei
  - Wuhan Puai Hosptial, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - Chenzhou No.1 People's Hospital, Chenzhou, Hunan
  - The First Affiliated Hospital Of University Of South China, Hengyang, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - Changzhou No.2 People's Hospital, Yanghu Branch, Changzhou, Jiangsu
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - Sir Run Run Hospital Nanjing Medical University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Jilin Province People's Hospital, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qinghai Provincial People's Hospital, Xining, Qinghai
  - The second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Jinan Central Hospital Affiliated to Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Qingdao Medical College, Qingdao, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Shanghai Pudong New Area People's Hospital, Pudong New District, Shanghai Municipality
  - Shanghai Huashan Hospital, Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji university, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hsopital, Tongji University, Shanghai, Shanghai Municipality
  - Dongfang Hospital Affiliated to Shanghai Tongji University, Shanghai, Shanghai Municipality
  - The Fifth People's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Tongren Hospital Shanghai Jiao Tong Univ. School of Medicine, Shanghai, Shanghai Municipality
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - First Affiated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The 2nd Affi Hosp of Zhejiang Univer School of Medicine, Hangzhou, Zhejiang
  - The Third Xiangya Hospital of Central South University, Changsha
- Czechia (5):
  - Nemocnice milosrdnych bratri, Brno
  - DIAMIN, Chrudim
  - Interna a diabetologie MUDr. Vodickova, Liberec
  - CCR Prague, Prague
  - MUDr. Michala Pelikanova, Prague
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- Romania (6):
  - SC Grand Med SRL, Oradea, Bihor County
  - S.C. Endodigest S.R.L., Oradea, Bihor County
  - SC Centru Medical Dr. Negrisanu SRL, Timișoara, Timiș County
  - SC Nutrilife SRL, Bucharest
  - Clinic of Diabetes Constanta, Constanța
  - Clinical County Emergency Hosp, Oradea
- Serbia (3):
  - Clinical Hospital Centre Dragisa Misovic, Belgrade
  - Endocrinology, Diabetes and Metabolism Diseases Clinic, Belgrade
  - Clinical Hospital Centre Zemun, Belgrade
- South Africa (10):
  - GCT, Arcadia, Gauteng
  - Dr R Dulabh, Johannesburg, Gauteng
  - Newtown Clinical Research, Johannesburg, Gauteng
  - WITS Clinical Research, Johannesburg, Gauteng
  - Clinresco Centres (Pty) Ltd, Kempton Park, Gauteng
  - Setshaba Research Centre, Soshanguve, Gauteng
  - Armansis Medical Centre, Brits, North West
  - Cape Town Medical Research Centre, Kuilsriver, Western Cape
  - Paarl Reserch Centre, Paarl, Western Cape
  - Union Hospital, Alberton
- Taiwan (4):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation - Linko Branch, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Derived] Ji L, Agesen RM, Bain SC, Fu F, Gabery S, Geng J, Li Y, Lu Y, Luo B, Pang W, Tao Y; PIONEER 12 investigators. Efficacy and safety of oral semaglutide vs sitagliptin in a predominantly Chinese population with type 2 diabetes uncontrolled with metformin: PIONEER 12, a double-blind, Phase IIIa, randomised trial. Diabetologia. 2024 Sep;67(9):1800-1816. doi: 10.1007/s00125-024-06133-4. Epub 2024 Jul 10. PMID 38985161

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 90 sites in 8 countries as follows: Brazil (3 sites), China (58 sites), Czech Republic (4 sites); Hong Kong (1 site), Romania (6 sites), Serbia (7 sites), Taiwan (4 sites), and South Africa (7 sites).
Pre-assignment Details: This was a 26-week, multicenter, multinational trial with four arms comparing efficacy and safety of oral semaglutide 3 milligram (mg), 7 mg and 14 mg once-daily with sitagliptin 100 mg once-daily. Out of 1441 participants randomized in the study, 1438 participants were exposed to trial product.
Groups:
- Oral Semaglutide 3 mg: Participants received semaglutide 3 mg tablet and placebo tablet matched to sitagliptin orally once daily for 26 weeks.
- Oral Semaglutide 7 mg: Participants received oral semaglutide tablets once daily in a dose escalation manner from week 0 to week 26: 3 mg from week 0 to week 4 and 7 mg from week 5 to week 26. Participants also received placebo matched to sitagliptin 100 mg for 26 weeks.
- Oral Semaglutide 14 mg: Participants received oral semaglutide tablets once daily in a dose escalation manner from week 0 to week 26: 3 mg from week 1 to week 4, 7 mg from week 5 to week 8 and 14 mg from week 9 to week 26. Participants also received placebo matched to sitagliptin 100 mg for 26 weeks.
- Sitagliptin 100 mg: Participants received oral sitagliptin 100 mg tablet and placebo tablet matched to oral semaglutide orally once daily for 26 weeks.
Period: Overall Study
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Started | 361 | 360 | 361 | 359
Full Analysis Set | 361 | 360 | 361 | 359
Safety Analysis Set | 361 | 358 | 361 | 358
Completed | 345 | 342 | 335 | 350
Not Completed | 16 | 18 | 26 | 9
Not completed — Withdrawal by Subject | 13 | 12 | 21 | 7
Not completed — Lost to Follow-up | 0 | 3 | 3 | 1
Not completed — Physician Decision | 1 | 1 | 1 | 1
Not completed — Death | 2 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg | Total
Number analyzed (Participants) | 361 | 360 | 361 | 359 | 1441
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (11.2) | 53.4 (10.8) | 53.5 (10.5) | 52.9 (10.9) | 53.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 147 | 146 | 156 | 601
  Male | 209 | 213 | 215 | 203 | 840
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 19 | 15 | 18 | 69
  Not Hispanic or Latino | 344 | 341 | 346 | 341 | 1372
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 272 | 270 | 271 | 271 | 1084
  Black or African American | 8 | 14 | 5 | 11 | 38
  NA | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Other | 8 | 11 | 18 | 18 | 55
  White | 73 | 65 | 67 | 59 | 264

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 26 in Glycated Haemoglobin (HbA1c) (%)
Description: Change in HbA1c from baseline to week 26 in percentage (%) point of HbA1c is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period and in-trial observation period. On-treatment without rescue medication observation period: from date of first dose of trial product following randomization and the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication. In-trial observation period: the time period where participants were considered to be in the trial, regardless of discontinuation of trial product or initiation of rescue medication.
Time Frame: From baseline to week 26
Population: Full analysis set (FAS) included all randomized participants. Overall Number of Participants Analyzed: participants with available data for this outcome measure and Number Analyzed: number of participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1C
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 344 | 340 | 332 | 350
Percentage point of HbA1C
  On-treatment observation period: number analyzed (Participants) | 321 | 315 | 298 | 334
  On-treatment observation period | -0.8 (1.0) | -1.3 (1.0) | -1.6 (1.0) | -0.7 (1.0)
  In-trial observation period | -0.8 (1.0) | -1.3 (1.0) | -1.5 (1.0) | -0.7 (1.0)
Statistical Analysis 1: Comparison: Oral Semaglutide 3 mg vs Sitagliptin 100 mg; Test type: Superiority; p = 0.0078, Mixed model for repeated measurements — Unadjusted two-sided p-value; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.3 to -0.1]
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg; Test type: Superiority; p < 0.0001, Mixed model for repeated measurements — Unadjusted two-sided p-value; Mean Difference (Net) = -0.7, 95% CI 2-sided [-0.8 to -0.6]
Statistical Analysis 3: Comparison: Oral Semaglutide 14 mg vs Sitagliptin 100 mg; Test type: Superiority; p < 0.0001, Mixed model for repeated measurements — Unadjusted two-sided p-value; Mean Difference (Net) = -1.0, 95% CI 2-sided [-1.1 to -0.8]

2. Secondary Outcome: Change From Baseline to Week 26 in Fasting Plasma Glucose (FPG)
Description: Change in fasting plasma glucose (FPG) from baseline to week 26 in millimole per liter (mmol/l) is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization and the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: From baseline to week 26
Population: FAS included all randomized participants. Overall Number of Participants Analyzed: participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 322 | 317 | 294 | 329
mmol/l | -1.03 (2.11) | -1.79 (2.20) | -2.00 (2.42) | -0.52 (2.36)

3. Secondary Outcome: Change From Baseline to Week 26 in Self-measured Plasma Glucose (SMPG) Profile: Mean 7-point Profile
Description: Change from baseline in mean 7-point SMPG profile at week 26 is presented. SMPG was recorded at the following 7 time points: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after dinner and at bedtime. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization and the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: From baseline to week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 300 | 311 | 290 | 317
mmol/L | -1.5 (2.2) | -2.3 (2.2) | -2.6 (2.2) | -1.2 (2.4)

4. Secondary Outcome: Change From Baseline to Week 26 in 7 Point SMPG Profile: Mean Postprandial Increment (Over All Meals)
Description: Change from baseline in 7-point SMPG: Mean postprandial increment (over all meals) at week 26 is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization and the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: From baseline to week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 301 | 311 | 290 | 317
mmol/L | -0.4 (2.0) | -0.9 (1.9) | -1.0 (2.1) | -0.6 (2.1)

5. Secondary Outcome: Number of Participants Who Achieved HbA1c <7.0 % (53 mmol/Mol) (American Diabetes Association [ADA] Target) (Yes/no)
Description: Number of participants who achieved HbA1c <7.0% (53 mmol/mol) (ADA target) is presented in category "Yes" and participants who could not achieve HbA1C <7.0 (53 mmol/mol) (ADA target) is presented in category "No". The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization and the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: At week 26
Population: FAS included all randomised participants. Overall Number of Participants Analyzed: participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 321 | 315 | 298 | 334
Participants
  Yes | 139 | 213 | 226 | 122
  No | 182 | 102 | 72 | 212

6. Secondary Outcome: Number of Participants Who Achieved HbA1c Equal to or Below 6.5 Percent (48 mmol/Mol) (American Association of Clinical Endocrinologists (AACE) Target) (Yes/no)
Description: Number of participants who achieved HbA1c equal to or below 6.5 percent (48 mmol/mol) (AACE target) (yes/no) is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization and the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: At week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 321 | 315 | 298 | 334
Participants
  Yes | 81 | 161 | 188 | 54
  No | 240 | 154 | 110 | 280

7. Secondary Outcome: Number of Participants Who Achieved HbA1c Reduction Equal to or Above 1 Percent-point (10.9 mmol/Mol) (Yes/no)
Description: Number of participants who achieved HbA1c reduction equal to or above 1 percent-point (10.9 mmol/mol) (yes/no) is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization and the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: At week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 321 | 314 | 298 | 334
Participants
  Yes | 141 | 203 | 226 | 129
  No | 180 | 111 | 72 | 205

8. Secondary Outcome: Time to Rescue Medication
Description: Time to rescue medication is presented as the number of participants who had taken rescue medication anytime from baseline to week 31. 'Rescue medication': use of new anti-diabetic medication as add-on to trial product and used for more than 21 days with the initiation at or after randomisation and before last day on trial product, and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before last day on trial product. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization and the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: From baseline to week 31
Population: FAS included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 361 | 360 | 361 | 359
Participants | 5 | 6 | 6 | 7

9. Secondary Outcome: Change From Baseline to Week 26 in Body Weight (Kilogram [kg])
Description: Change in body weight from baseline to week 26 in kg is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization and the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: From baseline to week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 322 | 319 | 300 | 335
Kilogram | -1.4 (3.0) | -2.9 (3.3) | -3.8 (3.7) | -0.5 (2.6)

10. Secondary Outcome: Percentage Change From Baseline to Week 26 in Body Weight
Description: Percentage change from baseline to week 26 in body weight is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization and the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: From baseline to week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 322 | 319 | 300 | 335
Percentage change | -2 (4) | -4 (4) | -5 (5) | -1 (3)

11. Secondary Outcome: Change From Baseline to Week 26 in Body Mass Index (BMI)
Description: Change from baseline in BMI is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization and the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: From baseline to week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 322 | 319 | 300 | 335
Kilogram per square meter (kg/m^2) | -0.5 (1.1) | -1.1 (1.2) | -1.4 (1.3) | -0.2 (0.9)

12. Secondary Outcome: Change From Baseline to Week 26 in Waist Circumference
Description: Change from baseline in waist circumference is presented. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization and the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: From baseline to week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 322 | 320 | 300 | 335
Centimeter | -1.6 (4.0) | -2.7 (4.4) | -3.7 (4.1) | -0.8 (3.4)

13. Secondary Outcome: Change From Baseline to Week 26 in Fasting Lipid Profile: Total Cholesterol (Ratio to Baseline)
Description: Change from baseline in total cholesterol (measured in mmol/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: From baseline to week 26
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 316 | 316 | 296 | 330
Ratio of total cholesterol | 1.00 (15.78) | 0.96 (17.34) | 0.96 (17.86) | 0.99 (19.69)

14. Secondary Outcome: Change From Baseline to Week 26 in Fasting Lipid Profile: Low-density Lipoprotein (LDL) Cholesterol (Ratio to Baseline)
Description: Change from baseline in LDL cholesterol (measured in mmol/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: From baseline to week 26
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 315 | 314 | 295 | 327
Ratio of LDL cholesterol | 1.02 (25.63) | 0.98 (28.70) | 0.98 (28.95) | 1.01 (30.12)

15. Secondary Outcome: Change From Baseline to Week 26 in Fasting Lipid Profile: Very-low-density Lipoprotein (VLDL) Cholesterol (Ratio to Baseline)
Description: Change from baseline in VLDL cholesterol (measured in mmol/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: From baseline to week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio of VLDL cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 315 | 315 | 295 | 327
Ratio of VLDL cholesterol | 1.05 (0.45) | 0.94 (0.37) | 0.94 (0.41) | 0.98 (0.43)

16. Secondary Outcome: Change From Baseline to Week 26 in Fasting Lipid Profile: High-density Lipoprotein (HDL) Cholesterol (Ratio to Baseline)
Description: Change from baseline in HDL Cholesterol (measured in mmol/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: From baseline to week 26
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 313 | 313 | 293 | 323
Ratio of HDL cholesterol | 1.02 (13.25) | 1.01 (14.42) | 1.00 (14.82) | 1.00 (16.03)

17. Secondary Outcome: Change From Baseline to Week 26 in Fasting Lipid Profile: Triglycerides (Ratio to Baseline)
Description: Change from baseline in triglycerides (measured in mmol/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: From baseline to week 26
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 315 | 315 | 295 | 327
Ratio of triglycerides | 0.96 (43.41) | 0.86 (46.28) | 0.86 (46.40) | 0.91 (44.29)

18. Secondary Outcome: Change From Baseline to Week 26 in Fasting Lipid Profile: Free Fatty Acids (Ratio to Baseline)
Description: Change from baseline in free fatty acids (measured in mmol/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to the end date which was the first date of any of the following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: From baseline to week 26
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of free fatty acids
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 308 | 308 | 290 | 318
Ratio of free fatty acids | 0.95 (56.36) | 0.89 (56.46) | 0.87 (66.18) | 0.96 (62.50)

19. Secondary Outcome: Change From Baseline to Week 26 in Short Form-36 Version 2 (SF-36v2) (Acute Version) Health Survey
Description: SF-36 v2.0 is a 36-item, patient-reported survey of patient health. SF-36 measures the participant's overall Health Related Quality of Life on 8 domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health) and two component summary scores (physical component summary and mental component summary). Range of score for domains and component summary scores : 1-100 (Higher scores indicated a better health state). A positive change score indicates an improvement since baseline. Outcome data was evaluated based on the on-treatment without rescue medication observation period: from date of first dose of trial product following randomization up to end date which was first date of any of following: the last dose of trial product plus 3 days or initiation of rescue medication.
Time Frame: From baseline to week 26
Population: FAS included all randomized participants. Overall Number of Participants Analyzed: participants with available data for this outcome measure and Number Analyzed: number of participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 322 | 320 | 299 | 334
Score on a scale
  Physical Function | 0.20 (5.63) | 0.48 (3.95) | 0.93 (4.51) | 0.31 (5.25)
  Role Physical | -0.47 (6.72) | -0.41 (6.82) | 0.28 (6.11) | 0.24 (7.27)
  Bodily Pain | -0.06 (8.44) | -0.37 (8.08) | 0.51 (8.03) | 0.22 (8.44)
  General Health | 1.47 (7.54) | 1.04 (7.09) | 1.95 (7.44) | 0.95 (7.19)
  Vitality | 0.44 (6.68) | 0.84 (6.64) | 1.21 (7.66) | 0.33 (7.28)
  Social Function | 0.49 (6.14) | -0.36 (6.45) | 0.17 (5.92) | 0.10 (6.36)
  Role Emotional | 0.06 (8.80) | -0.66 (8.37) | 0.23 (8.26) | 0.03 (8.40)
  Mental Health | 0.51 (7.01) | 0.33 (6.71) | 0.70 (7.34) | -0.7 (7.13)
  Physical Component | 0.15 (5.32) | 0.29 (4.74) | 0.98 (5.00) | 0.69 (5.62)
  Mental Component | 0.50 (6.71) | -0.07 (6.50) | 0.44 (6.75) | -0.39 (6.64)

20. Secondary Outcome: Number of Participants Who Achieved Body Weight Loss Equal to or Above 3 Percent (Yes/no)
Description: Number of participants who achieved body weight loss equal to or above 3 percent (yes/no) is presented. The outcome data was evaluated based on In-trial observation period: This observation period represented the time period where participants were considered to be in the trial, regardless of discontinuation of trial product or initiation of rescue medication. The in-trial observation period started at randomisation (as registered in the IWRS) and ended at the date of: The last direct participant-site contact, which was scheduled to take place 5 weeks after planned last dose of trial product at the follow-up visit; withdrawal for participants who withdrew their informed consent; The last participant-investigator contact as defined by the investigator for participants who were lost to follow-up; Death for participants who died before any of the above.
Time Frame: At week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 343 | 339 | 332 | 350
Participants
  Yes | 109 | 175 | 199 | 68
  No | 234 | 164 | 133 | 282

21. Secondary Outcome: Number of Participants Who Achieved Body Weight Loss Equal to or Above 5 Percent (Yes/no)
Description: Number of participants who achieved body weight loss equal to or above 5 percent (yes/no) is presented. The outcome data was evaluated based on In-trial observation period: This observation period represented the time period where participants were considered to be in the trial, regardless of discontinuation of trial product or initiation of rescue medication. The in-trial observation period started at randomisation (as registered in the IWRS) and ended at the date of: The last direct participant-site contact, which was scheduled to take place 5 weeks after planned last dose of trial product at the follow-up visit; withdrawal for participants who withdrew their informed consent; The last participant-investigator contact as defined by the investigator for participants who were lost to follow-up; Death for participants who died before any of the above.
Time Frame: At week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 343 | 342 | 333 | 351
Participants
  Yes | 55 | 107 | 149 | 28
  No | 288 | 235 | 184 | 323

22. Secondary Outcome: Number of Participants Who Achieved Body Weight Loss Equal to or Above 10 Percent (Yes/no)
Description: Number of participants who achieved body weight loss equal to or above 10 percent (yes/no). The outcome data was evaluated based on In-trial observation period: This observation period represented the time period where participants were considered to be in the trial, regardless of discontinuation of trial product or initiation of rescue medication. The in-trial observation period started at randomisation (as registered in the IWRS) and ended at the date of: The last direct participant-site contact, which was scheduled to take place 5 weeks after planned last dose of trial product at the follow-up visit; withdrawal for participants who withdrew their informed consent; The last participant-investigator contact as defined by the investigator for participants who were lost to follow-up; Death for participants who died before any of the above.
Time Frame: At week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 343 | 342 | 333 | 351
Participants
  Yes | 5 | 24 | 42 | 2
  No | 338 | 318 | 291 | 349

23. Secondary Outcome: Number of Participants Who Achieved HbA1c Below 7.0 Percent (53 mmol/Mol) Without Hypoglycaemia (Treatment-emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes) and no Body Weight Gain (Yes/no)
Description: Number of participants who achieved HbA1c < 7.0 percent (53 mmol/mol) without hypoglycaemia (treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes) and no body weight gain (yes/no) at week 26 is presented. The outcome data was evaluated based on In-trial observation period: This observation period represented the time period where participants were considered to be in the trial, regardless of discontinuation of trial product or initiation of rescue medication. The in-trial observation period started at randomisation (as registered in the IWRS) and ended at the date of: The last direct participant-site contact, which was scheduled to take place 5 weeks after planned last dose of trial product at the follow-up visit; withdrawal for participants who withdrew their informed consent; The last participant-investigator contact as defined by the investigator for participants who were lost to follow-up; Death for participants who died before any of the above.
Time Frame: At week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 344 | 339 | 332 | 350
Participants
  Yes | 114 | 195 | 222 | 79
  No | 230 | 144 | 110 | 271

24. Secondary Outcome: Number of Participants Who Achieved HbA1c Reduction Equal to or Above 1 Percent-point (10.9 mmol/Mol) and Body Weight Loss Equal to or Above 3 Percent (Yes/no)
Description: Number of participants who achieved HbA1c reduction equal to or above 1 percent-point (10.9 mmol/mol) and body weight loss equal to or above 3 percent (yes/no) is presented. The outcome data was evaluated based on In-trial observation period: This observation period represented the time period where participants were considered to be in the trial, regardless of discontinuation of trial product or initiation of rescue medication. The in-trial observation period started at randomisation (as registered in the IWRS) and ended at the date of: The last direct participant-site contact, which was scheduled to take place 5 weeks after planned last dose of trial product at the follow-up visit; withdrawal for participants who withdrew their informed consent; The last participant-investigator contact as defined by the investigator for participants who were lost to follow-up; Death for participants who died before any of the above.
Time Frame: At week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 344 | 339 | 332 | 350
Participants
  Yes | 64 | 128 | 159 | 33
  No | 280 | 211 | 173 | 317

25. Secondary Outcome: Number of Treatment-emergent Adverse Events During Exposure to Trial Product
Description: An adverse event (AE) was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. AEs with onset during the on-treatment period correspond to treatment-emergent AEs (TEAEs). The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 31
Population: Safety analysis set (SAS) included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 361 | 358 | 361 | 358
Events | 635 | 741 | 793 | 643

26. Secondary Outcome: Number of Treatment-emergent Severe or Blood Glucose Confirmed Symptomatic Hypoglycaemic Episodes During Exposure to Trial Product
Description: Number of treatment-emergent severe or blood glucose (BG) confirmed symptomatic hypoglycaemic episodes during exposure to trial product is presented. Severe: requiring assistance from another person for recovery. 'BG-confirmed': hypoglycaemic episode with a plasma glucose value < 3.1 mmol/L (56 mg/dL); The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 31
Population: SAS included all all participants exposed to at least one dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 361 | 358 | 361 | 358
Episodes | 2 | 2 | 2 | 1

27. Secondary Outcome: Change From Baseline to Week 26 in Haematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, and Neutrophils
Description: Change from baseline in hematology parameters such as basophils, eosinophils, lymphocytes, monocytes, and neutrophils were reported. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 26
Population: SAS included all participants exposed to at least one dose of trial product. Overall Number of Participants Analyzed: participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 310 | 305 | 290 | 320
10^9 cells per liter
  Basophils | 0.01 (0.05) | 0.01 (0.05) | 0.00 (0.04) | 0.00 (0.05)
  Eosinophils | 0.00 (0.11) | 0.00 (0.09) | -0.01 (0.25) | -0.00 (0.11)
  Lymphocytes | -0.03 (0.46) | 0.01 (0.40) | 0.00 (0.52) | 0.00 (0.39)
  Monocytes | 0.01 (0.15) | 0.01 (0.13) | 0.01 (0.14) | 0.02 (0.12)
  Neutrophils | 0.03 (1.08) | 0.13 (1.15) | 0.10 (1.22) | 0.31 (1.17)

28. Secondary Outcome: Change From Baseline to Week 26 in Haematology Parameter: Haematocrit (Ratio to Baseline)
Description: Change from baseline in Haematocrit at week 26 is reported as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 26
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of haematocrit
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 310 | 306 | 290 | 320
Ratio of haematocrit | 1.01 (6.76) | 1.00 (6.64) | 1.00 (6.21) | 1.00 (6.35)

29. Secondary Outcome: Change From Baseline to Week 26 in Haematology Parameter: Haemoglobin (Ratio to Baseline)
Description: Change from baseline in Haemoglobin at week 26 is reported as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 26
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of haemoglobin
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 310 | 306 | 290 | 320
Ratio of haemoglobin | 1.00 (5.71) | 1.00 (6.04) | 1.00 (5.47) | 1.00 (6.11)

30. Secondary Outcome: Change From Baseline to Week 26 in Haematology Parameter: Leucocytes (Ratio to Baseline)
Description: Change from baseline in Leucocytes at week 26 is reported as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 26
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of leucocytes
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 310 | 306 | 290 | 320
Ratio of leucocytes | 1.01 (19.28) | 1.02 (19.54) | 1.01 (21.24) | 1.04 (17.87)

31. Secondary Outcome: Change From Baseline to Week 26 in Haematology Parameter: Thrombocytes (Ratio to Baseline)
Description: Change from baseline in thrombocytes at week 26 is reported as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 26
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of thrombocytes
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 305 | 305 | 285 | 316
Ratio of thrombocytes | 0.99 (14.53) | 0.99 (16.65) | 0.99 (16.65) | 0.97 (15.65)

32. Secondary Outcome: Change From Baseline to Week 26 in Biochemistry Parameter: Calcium (Total) (Ratio to Baseline)
Description: Change from baseline in calcium (total) (measured in mmol/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 26
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of calcium
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 320 | 322 | 301 | 336
Ratio of calcium | 0.98 (4.40) | 0.98 (4.74) | 0.99 (4.80) | 0.98 (4.40)

33. Secondary Outcome: Change From Baseline to Week 26 in Biochemistry Parameter: Potassium (Ratio to Baseline)
Description: Change from baseline in potassium (measured in mmol/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 26
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of potassium
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 319 | 322 | 301 | 335
Ratio of potassium | 1.00 (8.51) | 1.00 (8.34) | 1.00 (8.96) | 1.01 (9.28)

34. Secondary Outcome: Change From Baseline to Week 26 in Biochemistry Parameter: Sodium (Ratio to Baseline)
Description: Change from baseline in sodium (measured in mmol/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 26
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of sodium
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 319 | 322 | 301 | 335
Ratio of sodium | 1.00 (1.58) | 1.00 (1.40) | 1.00 (1.49) | 1.00 (1.59)

35. Secondary Outcome: Change From Baseline to Week 26 in Biochemistry Parameter: Urea (Ratio to Baseline)
Description: Change from baseline in urea (measured in mmol/L) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 26
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of urea
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 320 | 322 | 301 | 336
Ratio of urea | 1.00 (26.29) | 0.99 (25.61) | 0.98 (23.78) | 1.03 (22.67)

36. Secondary Outcome: Change From Baseline to Week 26 in Biochemistry Parameter: Albumin (Ratio to Baseline)
Description: Change from baseline in Albumin (measured in grams per deciliter [g/dL]) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 26
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of albumin
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 320 | 323 | 303 | 337
Ratio of albumin | 0.99 (4.40) | 0.99 (4.57) | 0.99 (5.22) | 0.99 (5.05)

37. Secondary Outcome: Change From Baseline to Week 26 in Calcitonin (Ratio to Baseline)
Description: Change from baseline in calcitonin (measured in picograms per milliliter [pg/ml]) at week 26 is presented as ratio to baseline. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 26
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of calcitonin
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 324 | 324 | 301 | 335
Ratio of calcitonin | 1.00 (38.33) | 1.05 (35.56) | 1.02 (36.49) | 1.01 (31.96)

38. Secondary Outcome: Change From Baseline to Week 26 in Vital Signs: Pulse Rate
Description: Change from baseline in pulse rate is presented. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 26
Population: SAS included all participants exposed to at least one dose of trial product.
Measure: Mean (Standard Deviation); unit: Beats per minute (beats/min)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 361 | 358 | 361 | 358
Beats per minute (beats/min) | 78 (10) | 78 (11) | 78 (10) | 78 (10)

39. Secondary Outcome: Change From Baseline to Week 26 in Vital Signs: Systolic Blood Pressure
Description: Change from baseline in systolic blood pressure is presented. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 26
Population: SAS included all participants exposed to at least one dose of trial product.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 361 | 358 | 361 | 358
Millimeter of mercury (mmHg) | 131 (16) | 132 (15) | 130 (14) | 130 (14)

40. Secondary Outcome: Change From Baseline to Week 26 in Vital Signs: Diastolic Blood Pressure
Description: Change from baseline in diastolic blood pressure is presented. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 26
Population: SAS included all participants exposed to at least one dose of trial product.
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 361 | 358 | 361 | 358
Millimeter of mercury (mmHg) | 83 (10) | 84 (9) | 83 (10) | 83 (9)

41. Secondary Outcome: Change From Baseline to Week 26 in Electrocardiogram (ECG) Category
Description: Change from baseline in ECG category at week 26 is presented. Change from baseline results are presented as shift in findings categorized as: normal, abnormal and not clinically significant (NCS), and abnormal and clinically significant (CS). The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 26
Population: SAS included all participants exposed to at least one dose of trial product. Overall Number of Participants Analyzed: participants with available data for this outcome measure and Number Analyzed: number of participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 328 | 328 | 303 | 344
Participants
  Normal (Baseline) to normal (week 26): number analyzed (Participants) | 203 | 196 | 204 | 197
  Normal (Baseline) to normal (week 26) | 174 | 163 | 165 | 175
  Normal (Baseline) to abnormal NCS (week 26): number analyzed (Participants) | 203 | 196 | 204 | 197
  Normal (Baseline) to abnormal NCS (week 26) | 21 | 30 | 29 | 17
  Normal (Baseline) to abnormal CS (week 26): number analyzed (Participants) | 203 | 196 | 204 | 197
  Normal (Baseline) to abnormal CS (week 26) | 8 | 3 | 10 | 5
  Abnormal NCS (Baseline) to normal (week 26): number analyzed (Participants) | 85 | 91 | 71 | 109
  Abnormal NCS (Baseline) to normal (week 26) | 26 | 27 | 26 | 43
  Abnormal NCS (Baseline) to abnormal NCS (week 26): number analyzed (Participants) | 85 | 91 | 71 | 109
  Abnormal NCS (Baseline) to abnormal NCS (week 26) | 56 | 61 | 40 | 64
  Abnormal NCS (Baseline) to abnormal CS (week 26): number analyzed (Participants) | 85 | 91 | 71 | 109
  Abnormal NCS (Baseline) to abnormal CS (week 26) | 3 | 3 | 5 | 2
  Abnormal CS (Baseline) to normal (week 26): number analyzed (Participants) | 40 | 41 | 28 | 38
  Abnormal CS (Baseline) to normal (week 26) | 8 | 13 | 7 | 6
  Abnormal CS (Baseline) to abnormal NCS (week 26): number analyzed (Participants) | 40 | 41 | 28 | 38
  Abnormal CS (Baseline) to abnormal NCS (week 26) | 5 | 3 | 4 | 9
  Abnormal CS (Baseline) to abnormal CS (week 26): number analyzed (Participants) | 40 | 41 | 28 | 38
  Abnormal CS (Baseline) to abnormal CS (week 26) | 27 | 25 | 17 | 23

42. Secondary Outcome: Physical Examination Category
Description: The physical examination values for different body systems at baseline and week 26 are presented. The investigator interpreted the results and categorised them as: normal, abnormal NCS or abnormal CS. The physical examination are presented for the following body systems: cardiovascular system; central and peripheral nervous system; gastrointestinal system, including mouth; general appearance; head, ears, eyes, nose, throat, neck; lymph node palpation; musculoskeletal system; respiratory system; skin; and thyroid gland. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: Baseline and week 26
Population: SAS included all participants exposed to at least one dose of trial product. Number Analyzed: number of participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 361 | 358 | 361 | 358
Participants
  Cardiovascular system - Normal (Baseline) | 354 | 353 | 355 | 356
  Cardiovascular system - abnormal NCS (Baseline) | 5 | 4 | 6 | 2
  Cardiovascular system - Abnormal CS (Baseline) | 2 | 1 | 0 | 0
  Cardiovascular system -Normal (Week 26): number analyzed (Participants) | 327 | 326 | 305 | 341
  Cardiovascular system -Normal (Week 26) | 319 | 322 | 301 | 339
  Cardiovascular system - Abnormal NCS (Week 26): number analyzed (Participants) | 327 | 326 | 305 | 341
  Cardiovascular system - Abnormal NCS (Week 26) | 5 | 2 | 3 | 2
  Cardiovascular system - Abnormal CS (Week 26): number analyzed (Participants) | 327 | 326 | 305 | 341
  Cardiovascular system - Abnormal CS (Week 26) | 3 | 2 | 1 | 0
  Central and Peripheral Nervous System - Normal (Baseline) | 355 | 351 | 358 | 357
  Central and Peripheral Nervous System - Abnormal NCS (Baseline) | 2 | 5 | 3 | 1
  Central and Peripheral Nervous System - Abnormal CS (Baseline) | 4 | 2 | 0 | 0
  Central and Peripheral Nervous System - Normal (Week 26): number analyzed (Participants) | 326 | 326 | 305 | 341
  Central and Peripheral Nervous System - Normal (Week 26) | 322 | 321 | 302 | 339
  Central and Peripheral Nervous System - Abnormal NCS (Week 26): number analyzed (Participants) | 326 | 326 | 305 | 341
  Central and Peripheral Nervous System - Abnormal NCS (Week 26) | 2 | 3 | 2 | 2
  Central and Peripheral Nervous System - Abnormal CS (Week 26): number analyzed (Participants) | 326 | 326 | 305 | 341
  Central and Peripheral Nervous System - Abnormal CS (Week 26) | 2 | 2 | 1 | 0
  Gastrointestinal System incl. Mouth - Normal (Baseline) | 350 | 343 | 353 | 346
  Gastrointestinal System incl. Mouth - Abnormal NCS (Baseline) | 10 | 14 | 7 | 11
  Gastrointestinal System incl. Mouth - Abnormal CS (Baseline) | 1 | 1 | 1 | 1
  Gastrointestinal System incl. Mouth - Normal (Week 26): number analyzed (Participants) | 326 | 326 | 305 | 341
  Gastrointestinal System incl. Mouth - Normal (Week 26) | 314 | 315 | 300 | 329
  Gastrointestinal System incl. Mouth - Abnormal NCS (Week 26): number analyzed (Participants) | 326 | 326 | 305 | 341
  Gastrointestinal System incl. Mouth - Abnormal NCS (Week 26) | 12 | 10 | 4 | 10
  Gastrointestinal System incl. Mouth - Abnormal CS (Week 26): number analyzed (Participants) | 326 | 326 | 305 | 341
  Gastrointestinal System incl. Mouth - Abnormal CS (Week 26) | 0 | 1 | 1 | 2
  General Appearance - Normal (Baseline) | 329 | 325 | 328 | 328
  General Appearance - Abnormal NCS (Baseline) | 25 | 27 | 21 | 22
  General Appearance - Abnormal CS (Baseline) | 7 | 6 | 12 | 8
  General Appearance - Normal (Week 26): number analyzed (Participants) | 327 | 326 | 305 | 341
  General Appearance - Normal (Week 26) | 300 | 295 | 280 | 313
  General Appearance - Abnormal NCS (Week 26): number analyzed (Participants) | 327 | 326 | 305 | 341
  General Appearance - Abnormal NCS (Week 26) | 21 | 27 | 19 | 21
  General Appearance - Abnormal CS (Week 26): number analyzed (Participants) | 327 | 326 | 305 | 341
  General Appearance - Abnormal CS (Week 26) | 6 | 4 | 6 | 7
  Head, Ears, Eyes, Nose, Throat, Neck - Normal (Baseline): number analyzed (Participants) | 361 | 357 | 360 | 355
  Head, Ears, Eyes, Nose, Throat, Neck - Normal (Baseline) | 348 | 349 | 351 | 344
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal NCS (Baseline): number analyzed (Participants) | 361 | 357 | 360 | 355
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal NCS (Baseline) | 9 | 8 | 5 | 6
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal CS (Baseline): number analyzed (Participants) | 361 | 357 | 360 | 355
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal CS (Baseline) | 4 | 0 | 4 | 5
  Head, Ears, Eyes, Nose, Throat, Neck - Normal (Week 26): number analyzed (Participants) | 327 | 325 | 303 | 339
  Head, Ears, Eyes, Nose, Throat, Neck - Normal (Week 26) | 322 | 319 | 297 | 330
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal NCS (Week 26): number analyzed (Participants) | 327 | 325 | 303 | 339
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal NCS (Week 26) | 3 | 5 | 4 | 4
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal CS (Week 26): number analyzed (Participants) | 327 | 325 | 303 | 339
  Head, Ears, Eyes, Nose, Throat, Neck - Abnormal CS (Week 26) | 2 | 1 | 2 | 5
  Lymph Node Palpation - Normal (Baseline) | 361 | 353 | 357 | 357
  Lymph Node Palpation - Abnormal NCS (Baseline) | 0 | 5 | 3 | 1
  Lymph Node Palpation - Abnormal CS (Baseline) | 0 | 0 | 1 | 0
  Lymph Node Palpation - Normal (Week 26): number analyzed (Participants) | 326 | 326 | 305 | 341
  Lymph Node Palpation - Normal (Week 26) | 325 | 323 | 304 | 341
  Lymph Node Palpation - Abnormal NCS (Week 26): number analyzed (Participants) | 326 | 326 | 305 | 341
  Lymph Node Palpation - Abnormal NCS (Week 26) | 1 | 3 | 1 | 0
  Lymph Node Palpation - Abnormal CS (Week 26): number analyzed (Participants) | 326 | 326 | 305 | 341
  Lymph Node Palpation - Abnormal CS (Week 26) | 0 | 0 | 0 | 0
  Musculoskeletal System - Normal (Baseline) | 344 | 345 | 351 | 352
  Musculoskeletal System - Abnormal NCS (Baseline) | 13 | 8 | 7 | 4
  Musculoskeletal System - Abnormal CS (Baseline) | 4 | 5 | 3 | 2
  Musculoskeletal System - Normal (Week 26): number analyzed (Participants) | 326 | 326 | 305 | 341
  Musculoskeletal System - Normal (Week 26) | 314 | 319 | 301 | 335
  Musculoskeletal System - Abnormal NCS (Week 26): number analyzed (Participants) | 326 | 326 | 305 | 341
  Musculoskeletal System - Abnormal NCS (Week 26) | 6 | 4 | 2 | 3
  Musculoskeletal System - Abnormal CS (Week 26): number analyzed (Participants) | 326 | 326 | 305 | 341
  Musculoskeletal System - Abnormal CS (Week 26) | 6 | 3 | 2 | 3
  Respiratory System - Normal (Baseline) | 355 | 355 | 359 | 357
  Respiratory System -Abnormal NCS (Baseline) | 3 | 3 | 1 | 1
  Respiratory System - Abnormal CS (Baseline) | 3 | 0 | 1 | 0
  Respiratory System - Normal (Week 26): number analyzed (Participants) | 326 | 326 | 305 | 341
  Respiratory System - Normal (Week 26) | 324 | 325 | 305 | 341
  Respiratory System - Abnormal NCS (Week 26): number analyzed (Participants) | 326 | 326 | 305 | 341
  Respiratory System - Abnormal NCS (Week 26) | 2 | 1 | 0 | 0
  Respiratory System - Abnormal CS (Week 26): number analyzed (Participants) | 326 | 326 | 305 | 341
  Respiratory System - Abnormal CS (Week 26) | 0 | 0 | 0 | 0
  Skin - Normal (Baseline) | 282 | 282 | 296 | 277
  Skin - Abnormal NCS (Baseline) | 71 | 65 | 54 | 65
  Skin - Abnormal CS (Baseline) | 8 | 11 | 11 | 16
  Skin - Normal (Week 26): number analyzed (Participants) | 327 | 326 | 305 | 341
  Skin - Normal (Week 26) | 260 | 263 | 256 | 267
  Skin - Abnormal NCS (Week 26): number analyzed (Participants) | 327 | 326 | 305 | 341
  Skin - Abnormal NCS (Week 26) | 60 | 52 | 42 | 60
  Skin - Abnormal CS (Week 26): number analyzed (Participants) | 327 | 326 | 305 | 341
  Skin - Abnormal CS (Week 26) | 7 | 11 | 7 | 14
  Thyroid Gland - Normal (Baseline) | 356 | 351 | 358 | 350
  Thyroid Gland - Abnormal NCS (Baseline) | 4 | 4 | 1 | 4
  Thyroid Gland - Abnormal CS (Baseline) | 1 | 3 | 2 | 4
  Thyroid Gland - Normal (Week 26): number analyzed (Participants) | 327 | 326 | 305 | 341
  Thyroid Gland - Normal (Week 26) | 322 | 319 | 304 | 337
  Thyroid Gland - Abnormal NCS (Week 26): number analyzed (Participants) | 327 | 326 | 305 | 341
  Thyroid Gland - Abnormal NCS (Week 26) | 3 | 4 | 0 | 2
  Thyroid Gland - Abnormal CS (Week 26): number analyzed (Participants) | 327 | 326 | 305 | 341
  Thyroid Gland - Abnormal CS (Week 26) | 2 | 3 | 1 | 2

43. Secondary Outcome: Change From Baseline to Week 26 in Eye Examination Category
Description: The eye examination category at baseline and week 26 are presented. The investigator interpreted the results and categorised them as: normal, abnormal NCS or abnormal CS. The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 26
Population: as for outcome 42
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 361 | 358 | 361 | 358
Participants
  Left Eye Ophthalmoscopy - Normal (Baseline) | 245 | 240 | 254 | 248
  Left Eye Ophthalmoscopy - Abnormal NCS (Baseline) | 60 | 51 | 61 | 52
  Left Eye Ophthalmoscopy - Abnormal CS (Baseline) | 56 | 67 | 46 | 58
  Left Eye Ophthalmoscopy - Normal (Week 26): number analyzed (Participants) | 325 | 323 | 301 | 335
  Left Eye Ophthalmoscopy - Normal (Week 26) | 221 | 226 | 217 | 240
  Left Eye Ophthalmoscopy -Abnormal NCS (Week 26): number analyzed (Participants) | 325 | 323 | 301 | 335
  Left Eye Ophthalmoscopy -Abnormal NCS (Week 26) | 49 | 44 | 50 | 39
  Left Eye Ophthalmoscopy - Abnormal CS (Week 26): number analyzed (Participants) | 325 | 323 | 301 | 335
  Left Eye Ophthalmoscopy - Abnormal CS (Week 26) | 55 | 53 | 34 | 56
  Right Eye Ophthalmoscopy - Normal (Baseline): number analyzed (Participants) | 361 | 357 | 361 | 358
  Right Eye Ophthalmoscopy - Normal (Baseline) | 240 | 234 | 257 | 240
  Right Eye Ophthalmoscopy - Abnormal NCS (Baseline): number analyzed (Participants) | 361 | 357 | 361 | 358
  Right Eye Ophthalmoscopy - Abnormal NCS (Baseline) | 64 | 54 | 56 | 53
  Right Eye Ophthalmoscopy - Abnormal CS (Baseline): number analyzed (Participants) | 361 | 357 | 361 | 358
  Right Eye Ophthalmoscopy - Abnormal CS (Baseline) | 57 | 69 | 48 | 65
  Right Eye Ophthalmoscopy - Normal (Week 26): number analyzed (Participants) | 325 | 322 | 301 | 335
  Right Eye Ophthalmoscopy - Normal (Week 26) | 223 | 218 | 220 | 233
  Right Eye Ophthalmoscopy - Abnormal NCS (Week 26): number analyzed (Participants) | 325 | 322 | 301 | 335
  Right Eye Ophthalmoscopy - Abnormal NCS (Week 26) | 49 | 49 | 45 | 43
  Right Eye Ophthalmoscopy - Abnormal CS (Week 26): number analyzed (Participants) | 325 | 322 | 301 | 335
  Right Eye Ophthalmoscopy - Abnormal CS (Week 26) | 53 | 55 | 36 | 59

44. Secondary Outcome: Number of Participants With Treatment-emergent Severe or Blood Glucose Confirmed Symptomatic Hypoglycaemic Episodes During Exposure to Trial Product
Description: Number of participants with treatment-emergent severe or blood glucose (BG) confirmed symptomatic hypoglycaemic episodes during exposure to trial product is presented. Severe: requiring assistance from another person for recovery. 'BG-confirmed': hypoglycaemic episode with a plasma glucose value < 3.1 mmol/L (56 mg/dL); The outcome data was evaluated based on the on-treatment observation period: from date of first dose of trial product following randomization up to the first date of any of the following: follow-up visit, premature follow-up visit, last date on trial product plus 38 days or the end of the in-trial observation period.
Time Frame: From baseline to week 31
Population: SAS included all participants exposed to at least one dose of trial product.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 361 | 358 | 361 | 358
Participants | 2 | 2 | 2 | 1

ADVERSE EVENTS:
Time Frame: From baseline to week 31
Description: AEs with onset during the on-treatment period correspond to TEAEs. On-treatment observation period represented the time period where participants were considered treated with the trial product following randomization. Results are based on the SAS which included all participants exposed to at least one dose of trial product.
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Sitagliptin 100 mg
All-Cause Mortality (participants affected / at risk) | 2/361 | 2/358 | 1/361 | 0/358
Serious Adverse Events (participants affected / at risk) | 16/361 | 11/358 | 11/361 | 15/358
Other Adverse Events (participants affected / at risk) | 109/361 | 117/358 | 144/361 | 65/358
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 3 mg (N=361) | Oral Semaglutide 7 mg (N=358) | Oral Semaglutide 14 mg (N=361) | Sitagliptin 100 mg (N=358)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dacryocystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture treatment (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Keratitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimal gland abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 3 mg (N=361) | Oral Semaglutide 7 mg (N=358) | Oral Semaglutide 14 mg (N=361) | Sitagliptin 100 mg (N=358)
Decreased appetite (Metabolism and nutrition disorders) | 22 (22) | 30 (30) | 34 (39) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 30 (31) | 32 (40) | 48 (57) | 16 (17)
Lipase increased (Investigations) | 15 (15) | 17 (22) | 21 (23) | 12 (16)
Nausea (Gastrointestinal disorders) | 36 (38) | 39 (42) | 44 (50) | 14 (15)
Upper respiratory tract infection (Infections and infestations) | 26 (27) | 25 (29) | 31 (35) | 28 (35)
Vomiting (Gastrointestinal disorders) | 16 (17) | 18 (30) | 29 (38) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT04017832/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT04017832/SAP_001.pdf